CLINICAL TRIAL: NCT06062667
Title: Effect Of Fathers' Bırth Experıence On Paternal Attachment And Parentıng Perceptıon: A Randomızed Controlled Study
Brief Title: The Effect of Fathers' Birth Experience on Paternal Attachment and Parenting Perception: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Betul Uncu, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022/285
Record Dates: First submitted 2023-09-22; First posted 2023-10-02 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2023-10

CONDITIONS: Birth, First

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Fathers will accompany their husbands during the birth process
  Interventions: Other: accompany the birth
- Control group (No Intervention): routine maintenance

INTERVENTIONS:
Other: accompany the birth — Fathers will accompany their husbands during the birth process
  Arms: experimental group

SUMMARY:
In recent years, fathers have become increasingly involved in research, but research on fathers still lags behind research on mothers. During the transition to parenthood, a complex network of relationships emerges between father, mother and baby. During the process of becoming parents, mothers and fathers begin to bond with their unborn children. The prenatal period is hypothesized to be predictive of later postnatal attachment and perception of parenting. Paternal involvement at birth is associated with positive child health outcomes and parental well-being.

ELIGIBILITY:
Inclusion Criteria:

* Spouses of primiparous pregnant women who had spontaneous pregnancies and were admitted to the delivery room for normal labor were included in the study.

Exclusion Criteria:

* women without husbands

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Father
Enrollment: 100 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
The father-baby bonding of fathers who accompany their spouses in the delivery room is higher than fathers who do not accompany their spouses in the delivery room. | 15 days
  Primiparous pregnant women who had spontaneous pregnancies and were admitted to the delivery room for normal labor were included in the study. In determining the groups, participants were assigned to the Fathers Who Accompany the Birth (G1) and Fathers Who Did Not Accompany the Birth (G2) groups using web-based randomization (Randomizer.org). Pregnant women and their spouses in both groups who volunteered to participate in the study had the "Information Form" filled in after admission to the delivery room, and fathers filled out PAAQ and SPPRS. Two weeks after birth, the mother and father were contacted. PPAQ and SPPRS data were obtained from fathers and EPDS data were obtained from mothers.
  Information Form (IF), Paternal Antenatal Attachment Questionnaire (PAAQ), Self-Perception of Parental Role Scale (SPPRS), Postnatal Paternal-İnfant Attachment Questionnaire (PPAQ) Edinburg Postnatal Depression Scale (EPDS)

CONTACTS AND LOCATIONS:
Locations (1):
- Betül Uncu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No